CLINICAL TRIAL: NCT04792229
Title: Effects Of Whole Body Vibration On Lower Extremity With Diplegic Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC00821 Fatima Aslam
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Standing on WBV device (frequency of 40 Hz); 3 Minute vibration with 3 minute rest.
  Three times repetition . Total 18-minute vibrational therapy protocol. 3 days session per week
  Interventions: Other: Whole Body Viberation
- Control Group (Active Comparator): Stretching exercise (hip adductors ,plantar flexors, external rotators of hip & knee flexors).
  Active and passive ROMS to lower extremities. Strengthening exercises (hip and knee extensors, ankle dorsiflexes) 3 Repetitions into 3 day session per week
  Interventions: Other: Whole Body Viberation

INTERVENTIONS:
Other: Whole Body Viberation — WBV device (frequency of 40 Hz), 3 Minute vibration with 3 minute rest

SUMMARY:
This study will help to determine the beneficial effects of high frequency vibration on children with diplegic cerebral palsy in improving balance ,spasticity, strength of lower limb and quality of life and a comparison between the effect of simple conventional treatment and conventional management with the usage of vibrational therapy in cp patients.

DETAILED DESCRIPTION:
A study "Effect of whole body vibration training on mobility in children with cerebral palsy "states Whole body vibrational therapy induce an improvement in independent ambulation and mobility of lower limb by strengthening of muscles along with the refinement of walking pattern ,gait speed and stride length in children with cerebral palsy. On the basis of our study a better treatment protocol can be designed for future in diplegic spastic cerebral palsy children.

ELIGIBILITY:
Inclusion Criteria:

* Gross motor function classification level II-III
* Modified Ashworth Scale of 1-2

Exclusion Criteria:

* Auditory/ visually impaired
* Other neurological conditions e.g. spina bifida etc.
* Lower limb contractures
* Children with history of lower limb surgery in last 6 months

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 4 weeks
  the gold standard clinical tool, widely used for the measurement of the increased muscle tone and for grading the spasticity of the muscle. This scale is categorized in to 5 grades ranging from score 0 to 4. where 0 indicating normal muscular tone and 4 indicating marked spasticity of muscle. The intra class correlation coefficient for MAS is 0.92
Pediatric Balance Scale | 4 weeks
  an upgraded version of berg balance scale (inter-tester reliability of 0.997 and test-retest reliability of 0.9989) used for the assessment of the balance of school age children having mild to moderate level of developmental disorders , motor impairment or with brain lesion while performing functional activities

SECONDARY OUTCOMES:
Manual Muscle Testing | 4 weeks
  To assess the muscle strength, in clinical settings as well as in research trials evaluation done either manually with Manual Muscle Testing (MMT) or instrumentally by using a dynamometers .Inter-rater reliability of MMT is ICC 0.79-0.92)
CP QoL | 4 weeks
  Cp QOL have two versions :Primary caregiver (for parents of 4-12 aged children), composed of 65 items and Child self-report version (for children of 9-12 years of age ), 53 items questionnaire. Cp QOL (Caregiver ) is further Categorized into seven domains, Social wellbeing and acceptance, Participation and physical health, Feelings about functioning, Emotional wellbeing and self-esteem, Pain and impact of disability, Access to services, Family health.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, Principal Investigator — Riphah International University
Locations (1):
- Meshal School of Special Children, Tarbela, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No